CLINICAL TRIAL: NCT04089956
Title: Diaphragm Electrical Activity in "Spontaneous Breathing Challenge" Reliably Predict Early Extubation in Patients With Traumatic Cervical Spinal Cord Injury
Brief Title: EAdi as a Predictor of Successful Extubation in Patients With Traumatic Cervical Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Principal Investigator, Southeast University, China
Other Study IDs: 20190911
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Traumatic Cervical Spinal Cord Injury (CSCI)
Keywords: spinal cord injury; weaning
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extubation Success: extubation Success which defined as no need of reintubation or tracheostomy after extubation.
  Interventions: Other: No interventation
- Extubation Failure: Extubation Failure was defined as need for any invasive ventilatory support after fist extubation during ICU stay or tracheostomy befor any extubation attempt.
  Interventions: Other: No interventation

INTERVENTIONS:
Other: No interventation — A retrospective cohort Observational study with no intervention

SUMMARY:
Esophageal recordings of diaphragm electrical activity (EAdi) made it possible to monitor respiratory drive and the subsequent phrenic nerve conduction and respiratory neuromuscular function continuously. Thus, we designed a "spontaneous breathing challenge" test to monitor the change in EAdi after a maximal inspiration. We hypothesized that the absolute change (ΔEAdi) and the percentage changes change (ΔEAdi%) in EAdi after a "spontaneous breathing challenge" predict successful extubation in traumatic CSCI patients during acute hospitalization.

DETAILED DESCRIPTION:
A retrospective cohort study enrolled adult traumatic CSCI patients who underwent mechanical ventilation and admitted to the intensive care unit (ICU) of Zhongda hospital form June 2014 to July 2018. The following inclusion criteria were used: age 18 years or older, traumatic CSCI patients with a neurologic level of injury of C1 to C8 by the American Spinal Injury Association (ASIA) standard impairment scale grade A-D patients with mechanical ventilation due to acute respiratory failure and admite to ICU, dedicated nasogastric tube with nine electrodes that allow to continuously measure diaphragm electrical activity (EAdi catheter, Maquet, Solna, Sweden) in postion. CSCI was defined as radiologically-confirmed injury to the cervical spinal column, combined with clinical signs and symptoms consistent with CSCI at that level. The exclusion criteria were: tracheostomy at time of addmition to ICU, withhold or withdraw life sustaining treatment due to other serious organ injury, can't complete instructional actions, death occurred within 7 days after injury, or postoperative MV was a direct result of surgery and had duration of less than 24 hours postoperatively. Extubation or tracheostomy was decided by the physician in charge according to the local protocol of weaning.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older
2. Traumatic CSCI patients with a neurologic level of injury of C1 to C8 by the American Spinal Injury Association (ASIA) standard impairment scale grade A to D
3. patients with mechanical ventilation due to acute respiratory failure and admit to ICU
4. with dedicated nasogastric tube with nine electrodes that allow to continuously measure diaphragm electrical activity (EAdi catheter, Maquet, Solna, Sweden) in position.

Exclusion Criteria:

1. tracheostomy before ICU admission
2. withhold or withdraw life sustaining treatment due to other serious organ injury
3. can't complete instructional actions,
4. death occurred within 7 days after injury
5. postoperative MV was a direct result of surgery and had duration of less than 24 hours postoperatively.
6. EAdi data not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Traumatic CSCI patients with mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
extubation Success | up to 90 days
  defined as no reintubation after first extubation and no tracheostomy before any extubation attempt during ICU stay

SECONDARY OUTCOMES:
ventilator free days | up to 28 days
  days of nowvntilation at day 7,14,28
complications | up to 90 days
  complications of mechanication ventilation such as VAP and so on
mortality | up to 90 days
  in-ICU and in hospital mortality
length of stay | up to 90 days
  length of stay in-ICU and in hospital

CONTACTS AND LOCATIONS:
Overall Officials: LING LIU, Study Director — Zhongda Hospital
Locations (1):
- Ling Liu, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided